CLINICAL TRIAL: NCT03605459
Title: Validation Study: A Prospective, Non-Randomized, Single Arm Trial to Assess the Efficacy of the Comfort Plug™ in Preventing Urinary Incontinence in Male Subjects With Post Prostatectomy Urinary Incontinence (COMFORT STUDY)
Brief Title: Trial to Assess the Efficacy of the Comfort Plug™in Preventing Urinary Incontinence (COMFORT STUDY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMX Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX-UR-2013-004
Record Dates: First submitted 2014-02-07; First posted 2018-07-30 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device use (Experimental): Only one treatment arm; the "Comfort Plug™" is a device designed to control urinary incontinence in male subjects by being placed in the urethra to stop urine leakage.
  Interventions: Device: Comfort Plug™

INTERVENTIONS:
Device: Comfort Plug™

SUMMARY:
Validation Study: A Prospective, Non-Randomized, Single Arm Trial to Assess the Efficacy of the Comfort Plug™ in Preventing Urinary Incontinence in Male Subjects with Post Prostatectomy Urinary Incontinence (COMFORT STUDY)

DETAILED DESCRIPTION:
This is a first-in-human, device assessment, feasibility study to assess the safety, effectiveness, comfort and usability of the prototype Comfort Plug™ for controlling urinary incontinence in male subjects. No drug treatment will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Male 18 years of age or older
2. At least 6 months post radical prostatectomy for localized prostate cancer
3. Cystoscopic evaluation of the lower urinary tract within 12 months of screening
4. Eastern Cooperative Oncology Group (ECOG) 0 or 1 performance status
5. Evidence of moderate to severe urinary incontinence as assessed by the investigator, requiring protective garments or pads
6. Post-surgical Prostate Specific Antigen (PSA) <0.04

Exclusion Criteria:

1. Inability to insert the Comfort Plug™ into his own urethra and remove it
2. History of significant incontinence prior to radical prostatectomy
3. Evidence of incomplete bladder emptying post radical prostatectomy
4. Recurrent , refractory bacteruria
5. Urethral stricture disease.
6. History of meatal stenosis or phimosis
7. History of any other malignancy except basal cell skin cancer
8. Planned radiotherapy for post prostatectomy residual disease within the next 90 days
9. Evidence of neurogenic bladder dysfunction
10. Multiple sclerosis or previous spinal cord trauma/pathology resulting in any neurologic deficit that, in the opinion of the investigator, might compromise the outcome
11. Ongoing constipation
12. Use of anticoagulant or antiplatelet medications excluding low-dose Acetylsalicylic acid (ASA)
13. Hemophilia
14. Any cardiac condition that requires the use of pre-procedure antibiotic prophylaxis such as a mechanical valve
15. Currently receiving successful medical treatment for incontinence.
16. The usage of male urethral slings
17. Planning to travel by airplane during the course of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
To establish safety of the Comfort Plug | 30 days
  Safety is characterized by the absence of complications and adverse events
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | 30 days
  The ICIQ is a psychometrically robust patient-completed questionnaire for evaluating the frequency, severity and impact of urinary incontinence (UI) on Quality of Life in men and women. The ICIQ-SF is scored from 0 to 21, with greater scores indicating increased severity of UI. The change from baseline (Visit Day 0) in the ICIQ-SF score at Visit Days 7 and 30 (cohort 1) or Visit Days 14 and 30 (subsequent cohorts) will be examined.
Weight of protective pads | 30 days
  Change from baseline (Visit Day 0) in the weight of the protective pads a Visit Days 7 and 30 (cohort 1) or Visit Days 14 and 30 (subsequent cohorts).

SECONDARY OUTCOMES:
Incontinence Quality of Life Questionnaire (I-QOL) | 30 days
  The questionnaire has a scale of 22-110; The higher the score, the less incontinence is having a negative impact on the subject's Quality of Life. Change from baseline (Visit Day 0) in the I-QOL instrument scores at Visit Days 14 and 30 for i) avoidance and limiting behavior ii) psychosocial impacts iii) social embarrassment will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Casey, MD, Study Director — CMX Research
Locations (4):
- Canada (4):
  - Southern Interior Medical Research, Kelowna, British Columbia
  - The Fe/Male Health Centres, Oakville, Ontario
  - 643094 Ontario Inc., Scarborough Village, Ontario
  - Dr. Dean Elterman Medicine Professional Corporation, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Abstract from the CUAJ June 2020 (page S59 & S60) — https://cuaj.ca/index.php/journal/article/view/6732/4463